CLINICAL TRIAL: NCT04849871
Title: Evaluation of Single Fraction Accelerated Partial Breast Irradiation vs. Five Fraction Accelerated Partial Breast Irradiation for Low-risk Stage 0 and I Breast Carcinoma - BreaStBRT
Brief Title: Single Fraction Accelerated Partial Breast Irradiation vs. Five Fraction Accelerated Partial Breast Irradiation for Low-risk Stage 0 and I Breast Carcinoma
Acronym: BreaStBRT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202104085
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma; Breast Cancer; Stage 0 Breast Cancer; Stage I Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm S_APBI (External Beam Accelerated Partial Breast Irradiation (APBI) 20 Gy-1 fraction) (Experimental): -External Beam APBI 20 Gy to surgical bed surface (7 Gy to 1 cm from surgical bed in 1 fraction)
  Interventions: Radiation: External Beam Accelerated Partial Breast Irradiation
- Arm F_APBI (External Beam Accelerated Partial Breast Irradiation (APBI) 30 Gy-5 fractions) (Experimental): -External Beam APBI 30 Gy in 5 fractions over 5 days.
  Interventions: Radiation: External Beam Accelerated Partial Breast Irradiation

INTERVENTIONS:
Radiation: External Beam Accelerated Partial Breast Irradiation — APBI simulation must take place no more than 8 weeks from final definitive breast surgery.
  Other Names: APBI

SUMMARY:
This study will evaluate the local control, complication rates, cosmetic results, and quality of life between patients treated with a single fraction vs. five fractions of accelerated partial breast irradiation (S_APBI vs. F_APBI) when used as the sole method of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* AJCC 7th Edition stage 0 or I (TisN0 ≤ 2 cm or T1N0) histologically confirmed carcinoma of the breast, treated with partial mastectomy. Axillary sampling is required only for cases of invasive cancers. Tumor size is determined by the pathologist. Clinical size may be used if the pathologic size is indeterminate. Patients with invasive cancer must have no positive axillary lymph nodes with at least 6 axillary lymph nodes as assessed by axillary ultrasound, axillary sampling, or axillary sentinel node procedure.
* Negative histologic margins of partial mastectomy or re-excision specimen. The posterior margin is always considered widely negative if the partial mastectomy extended to the pectoralis fascia and there is no tumor on ink. Margins generally are positive if there is invasive or noninvasive tumor at the inked resection margin, close but negative if the tumor is within 2 mm of the inked margin and negative if the tumor is at least 2 mm away from the inked edge.[42]
* Invasive ductal, lobular, medullary, papillary, colloid (mucinous), tubular histologies, or mixed histologies (lesions ≤ 2 cm) that are estrogen and/or progesterone receptor positive and do not exhibit HER2/neu gene amplification OR ductal carcinoma in situ (lesions ≤ 2 cm) that are estrogen and/or progesterone receptor positive.
* Neoadjuvant hormone therapy, chemotherapy, or biologic therapy is not allowed prior to APBI, but adjuvant hormone therapy may have been started after surgery. Planned chemotherapy or biologic therapy must not start for at least 4 weeks after the completion of APBI.
* Good candidate for treatment per protocol in the judgment of the PI and/or treating physician following simulation.
* Postmenopausal status.
* Age ≥ 50 years at diagnosis.
* Able to understand and willing to sign IRB-approved written informed consent document.
* All radiation therapy must be planned for delivery at BJH or a BJH/Siteman satellite location with the following stipulations: F_APBI may be delivered at any Siteman location. S_APBI treatment must occur at the main Siteman location at BJH and will be delivered on a Viewray Unit, the Varian Edge unit, or the Varian Halcyon unit. Pre and post treatment care is allowed at any Siteman center.

Exclusion Criteria:

* Presence of distant metastases.
* Nonepithelial breast malignancies such as sarcoma or lymphoma.
* Proven multicentric carcinoma (tumors in different quadrants of the breast, or tumors separated by at least 4 cm) with other clinically or radiographically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy.
* Histologically confirmed positive axillary nodes in the ipsilateral axilla. Palpable or radiographically suspicious contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor.
* Prior non-hormonal therapy for the present breast cancer, including radiation therapy or chemotherapy.
* Diagnosis of systemic lupus erythematosis, scleroderma, or dermatomyositis.
* Diagnosis of a coexisting medical condition which limits life expectancy to < 2 years.
* Paget's disease of the nipple.
* Skin involvement, regardless of tumor size.
* Unsatisfactory breast for APBI as determined by the treating physician. For example, if there is little breast tissue remaining between the skin and pectoralis muscle after surgery, treatment with APBI is technically problematic.
* Partial mastectomy so extensive that the cosmetic result is fair or poor prior to APBI as determined by the treating physician.
* Surgical margins which cannot be microscopically assessed or are positive at pathological evaluation.
* Time between final definitive breast surgical procedures to APBI simulation is greater than 8 weeks.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2029-08-06 (Estimated); Study Completion 2029-08-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are free of breast cancer in the treated breast (IBTR) | Through 5 years after completion of treatment (estimated to be 5 years and 5 days)
  -IBTRs will be categorized as local (infield) if they occur within the prescription isodose volume, peripheral if between the prescription isodose volume and a volume 2 cm outside of the prescription isodose volume, and non-contiguous or extrafield if they are beyond the peripheral volume described above.
Feasibility of treatment regimen as measured by the ability to complete accrual to the trial in 3 years | Through enrollment of all participants (estimated to be 3 years)

SECONDARY OUTCOMES:
Proportion of patients who are free of breast cancer in the regional lymph nodes | Through 5 years after completion of treatment (estimated to be 5 years and 5 days)
  -Regional lymph nodes are ipsilateral axilla, infraclavicular, supraclavicular, and internal mammary groups.
Proportion of patients who are free of distant disease | Through 5 years after completion of treatment (estimated to be 5 years and 5 days)
Proportion of patients who are alive | Through 5 years after completion of treatment (estimated to be 5 years and 5 days)
Change in quality of life as measured by EORTC QLQ-C30 | Baseline, 6 months post-end of radiation therapy (RT), 12 months post-end of RT, 24 months post-end of RT, 36 months post-end of RT, 4 years post-end of RT, and 5 years post-end of RT
  * The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  * All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Change in quality of life as measured by EORTC QLQ-BR23 | Baseline, 6 months post-end of radiation therapy (RT), 12 months post-end of RT, 24 months post-end of RT, 36 months post-end of RT, 4 years post-end of RT, and 5 years post-end of RT
  * The QLQ-BR23 is a breast-specific module that comprises of 23 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss.
  * All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Change in cosmesis as measured quantitatively by the Breast Retraction Assessment (BRA) | Before treatment, 4-8 month follow-up, 10-14 month follow-up, 2 years, 3 years, 4 years, and 5 years (estimated to be 5 years)
  -Breast Retraction Assessment (BRA) is an objective evaluation of the amount of cosmetic retraction of the treated breast in comparison to the untreated breast in patients. A clear acrylic sheet supported vertically and marked as a grid at 1 cm intervals is employed to perform the measurements.
Change in cosmesis as measured quantitatively by the Percent Breast Retraction Assessment (pBRA) | Before treatment, 4-8 month follow-up, 10-14 month follow-up, 2 years, 3 years, 4 years, and 5 years (estimated to be 5 years
  -Breast Retraction Assessment (BRA) is an objective evaluation of the amount of cosmetic retraction of the treated breast in comparison to the untreated breast in patients. A clear acrylic sheet supported vertically and marked as a grid at 1 cm intervals is employed to perform the measurements.
Change in cosmesis as measured qualitatively by the Aronson modified Harris scale (physician graded) | Before treatment, 4-8 month follow-up, 10-14 month follow-up, 2 years, 3 years, 4 years, and 5 years (estimated to be 5 years
  -The following general descriptors will be used:
  * Excellent - when compared to the untreated breast, there is minimal or no difference in the size, shape, or texture of the treated breast. There may be mild thickening or scar tissue within the breast or skin, but not enough to change the appearance.
  * Good - there is mild asymmetry in the size or shape of the treated breast as compared to the normal breast. The thickening or scar tissue within the breast causes only a mild change in the shape.
  * Fair - there is obvious difference in the size and shape of the treated breast. This change involves ¼ or less of the breast.
  * Poor - marked change in the appearance of the treated breast involving more than ¼ of the breast tissue.
Change in cosmesis as measured qualitatively by the Aronson modified Harris scale (patient graded) | Before treatment, 4-8 month follow-up, 10-14 month follow-up, 2 years, 3 years, 4 years, and 5 years (estimated to be 5 years
  -The following general descriptors will be used:
  * Excellent - when compared to the untreated breast, there is minimal or no difference in the size, shape, or texture of the treated breast. There may be mild thickening or scar tissue within the breast or skin, but not enough to change the appearance.
  * Good - there is mild asymmetry in the size or shape of the treated breast as compared to the normal breast. The thickening or scar tissue within the breast causes only a mild change in the shape.
  * Fair - there is obvious difference in the size and shape of the treated breast. This change involves ¼ or less of the breast.
  * Poor - marked change in the appearance of the treated breast involving more than ¼ of the breast tissue.
Presence of complications | From start of treatment through 5 years (estimated to be 5 years and 5 days)
Occurrence of mastectomy after completion of initial breast-conserving treatment | Through 5 years after completion of treatment (estimated to be 5 years and 5 days)
Frequency of any CTCAE v5.0 grade 3-4 toxicities | From start of treatment through 5 years (estimated to be 5 years and 5 days)
Proportion of patients who are free of acute serious treatment related toxicity | From start of treatment until 6 months post-treatment (estimated to be 6 months)
  * Serious treatment related toxicity are those treatment-related grade 3 or higher adverse events as measured by CTCAE v5.0
  * Toxicities of concern include breast pain, delayed wound healing, persistent seroma fluid accumulation, breast fibrosis, and fat necrosis in the treated breast. Rare toxicities include radiation pneumonitis, coronary artery disease, and pericarditis.
Proportion of patients who are free of late serious treatment related toxicity | From 6 months through 5 years (estimated to be 4.5 years)
  * Serious treatment related toxicity are those treatment-related grade 3 or higher adverse events as measured by CTCAE v5.0
  * Toxicities of concern include breast pain, delayed wound healing, persistent seroma fluid accumulation, breast fibrosis, and fat necrosis in the treated breast. Rare toxicities include radiation pneumonitis, coronary artery disease, and pericarditis.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Zoberi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu